CLINICAL TRIAL: NCT05601531
Title: Extraction Socket Sealed with Autologous Tooth Root in Ridge Preservation
Brief Title: Autologous Tooth Root in Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiang-Hsi Hong, Professor-level attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202002350A0
Record Dates: First submitted 2022-10-21; First posted 2022-11-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-11

CONDITIONS: Alveolar Ridge Preservation
MeSH Terms: interventions — Calcitriol; Bone Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Autologous Tooth Root+Vit.D3+Bone graft (Experimental): Placement of bone graft and local administration of Vit.D3, and placement of autologous root slices
  Interventions: Procedure: Autologous Tooth Root; Drug: Vit.D3; Other: bone graft
- Autologous Tooth Root+ Bone graft (Experimental): Placement of bone graft without local administration of Vit.D3 and placement of autogenous root slices
  Interventions: Procedure: Autologous Tooth Root; Other: bone graft
- Bone graft (Experimental): Only bone graft materials were placed, no local administration of Vit.D3, and no autologous root slices were placed
  Interventions: Other: bone graft
- Natural healing (No Intervention): After the wound healed naturally, no bone graft material was filled, and Vit.D3 was not administered locally, and autologous tooth root slices were not placed.

INTERVENTIONS:
Procedure: Autologous Tooth Root — An autologous Tooth Root is made from one's own tooth root and covered in an extraction socket where bone graft is placed.
  Arms: Autologous Tooth Root+ Bone graft; Autologous Tooth Root+Vit.D3+Bone graft
Drug: Vit.D3 — Local administration of Vit.D3, through the effect of Vit.D3 to explore whether it can help to accelerate the healing of tooth extraction cavity and the clinical effectiveness of bone regeneration.
  Other Names: calcitriol
  Arms: Autologous Tooth Root+Vit.D3+Bone graft
Other: bone graft — Selecting bone materials for alveolar ridge preservation according to treatment needs
  Other Names: BG
  Arms: Autologous Tooth Root+ Bone graft; Autologous Tooth Root+Vit.D3+Bone graft; Bone graft

SUMMARY:
Use your extracted teeth for routine dental care to make an autologous root slice, cover it in your extraction cavity, and give you Vit.D3 locally with the bone material you use. The difference from traditional therapy is autologous Local use of tooth root slices and Vit.D3, bone materials and Vit.D3 are already qualified drugs on the market, but there is no precedent for making slices from autologous tooth roots, which will be a new medical technology that has not been used before test.

DETAILED DESCRIPTION:
The anatomy of the alveolar bone around the teeth can be altered by tooth extraction. Bone ridge preservation can preserve/improve the quality and quantity of alveolar bone for future implants or dentures to promote predictable function and esthetics; in addition, extraction cavity closure can be used as an aid, in vertical or alveolar ridges. Horizontal preservation had significantly better clinical outcomes. According to the treatment needs, appropriate bone materials were selected for bone ridge preservation and local administration of Vit.D3, and the extraction cavity closure was performed with autologous root slices to observe and track the therapeutic effect. Free gingival grafts or pedicle soft tissue grafts can help bone and spine preservation with good clinical outcomes, but autologous soft tissue grafts can increase wounds at the donor site and increase the patient's postoperative discomfort. Collagen sponges can help bone graft materials. Stay in the extraction cavity, promote the formation and fixation of blood clots, and prevent soft tissue from growing in, but collagen degrades rapidly, and it will decompose faster once the nearby tissue has symptoms of acute inflammation. The advantage of autologous root slices is that it is biocompatible High performance, it can effectively isolate the bone graft material from the contamination of the oral environment, and it will not absorb or be infected due to the acute inflammation of the nearby tissue. Wounds can reduce postoperative discomfort, so the use of autologous tooth root slices without the periodontal ligament exposed to the oral environment is less likely to cause infection or premature absorption, and can effectively protect the stability of blood clots in the extraction cavity. , reduce the saliva contamination of bone graft materials, and at the same time will not increase the cost of materials or the economic burden of the patient, the side with the periodontal ligament can also promote bone formation and help the retention of alveolar bone, which is both novel and good. The method of sealing the extraction socket can improve the predictability and aesthetics of the bone and spine preservation surgery, and help the patient to be replanted in an ideal position in the future. It is also hoped that the effect of Vit.D3 in promoting bone regeneration can accelerate the healing of the extraction socket.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign written subject consent to surgery
2. The extraction socket is located in the anterior and posterior areas of the upper and lower jaws.
3. The intraoral extraction socket (bone defect) area will need to receive artificial dental implant treatment in the future.
4. The patient does not have systemic disease.
5. Patients who do not have systemic diseases (such as hypertension, diabetes, heart disease, osteoporosis, bone-related diseases, kidney diseases, thyroid and parathyroid diseases, etc.), and those who need to take preventive antibiotics before tooth extraction/surgery (artificial valve/stent, artificial joint).

Exclusion Criteria:

1. Patients with potentially impaired healing capacity such as cancer, diabetes, bone infection, tuberculosis, hemoglobin abnormal anemia or congenital immunodeficiency conditions, cellulitis, acute periodontal cysts, severe cusp lesions (cyst size) >2mm2) or subjects with dental and jaw lesions.
2. Women who are pregnant or breastfeeding.
3. Exclude heavy smokers or betel nut chewers who smoke more than one pack of cigarettes per day.
4. The bone defect of the extraction socket is severe (especially if the vertical height of the buccal bone defect [corono-apical] exceeds 1/2), other bone regeneration surgery (GBR) is required, otherwise it is impossible to have sufficient alveolar bone height in the future and widths to provide artificial dental implants
5. The root of the tooth has been severely damaged, the root of the active periodontal ligament is lacking, and it is not suitable for autologous root sectioning, and the alveolar bone and apical defect after tooth extraction are severe (the apical lesion with a defect diameter of >3mm in root apex X-ray examination) [apical lesion])

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline 3D computed tomography data at 12th~16th week | At the 12th~16th week of the experiment
  This experiment mainly used the relative position of the extraction socket and the adjacent tooth CEJ in CT images for height positioning and correction, and measured and compared the changes of the width and height of the bone ridge and the shape and volume during the treatment. The Hu value of the adjacent dentin of the secondary CT was used as the standard and correction to measure and compare the change of the Hu value of the extraction socket during the treatment
Change from baseline X-ray apical film data at 12th~16th week | At the 12th~16th week of the experiment
  Irradiate X-rays before implantation or other treatment operations, record the width and height of the alveolar bone and the relative position to the CEJ of the adjacent teeth, and compare the pixel values between the extraction socket and the adjacent non-extraction area. By calculating the number of images The difference of pixel values before and after tooth extraction healing can be inferred by judging the gray-scale depth (ie density) of the image.
Tissue Section Analysis | Average 12th~16th week of the experiment, the day of implant surgery
  During artificial dental implant surgery, 3mm diameter x 6mm depth alveolar bone was taken out for section observation. Hematoxylin and eosin staining (H&E) was used to observe the morphology of bone tissue. At the same time, the sections were subjected to immunohistochemical staining (IHC) to observe bone-related biomarkers, and optical microscopy was used to perform morphological analysis and to analyze the difference in the rate of new bone formation.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang H Hong, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No